CLINICAL TRIAL: NCT00118196
Title: A Phase II Study of Arsenic Trioxide in Combination With 5-Azacitidine in Myelodysplastic Syndromes
Brief Title: Azacitidine and Arsenic Trioxide in Treating Patients With Myelodysplastic Syndromes or Chronic Myelomonocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to limited resources available to conduct study
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000433313; MUSC-MDS2773; MUSC-15348
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; chronic myelomonocytic leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Arsenic Trioxide; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: arsenic trioxide
Drug: azacitidine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as azacitidine and arsenic trioxide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving azacitidine together with arsenic trioxide works in treating patients with myelodysplastic syndromes or chronic myelomonocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with myelodysplastic syndromes or chronic myelomonocytic leukemia treated with azacitidine and arsenic trioxide.

Secondary

* Determine time to treatment failure in patients treated with this regimen.
* Determine the tolerability and toxicity of this regimen in these patients.
* Determine progression-free survival of patients treated with this regimen.

OUTLINE: This a multicenter, non-randomized, open-label, study.

Patients receive azacitidine subcutaneously once daily on days 1-5 and arsenic trioxide IV over 1-2 hours on days 1, 2, 8, 9, 15, 16, 22, and 23. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are evaluated for response on day 113 (week 17). Patients with disease progression or no response are removed from the study. Patients achieving a complete response (CR) receive 2 additional courses of therapy and then undergo observation. Patients achieving a partial response receive 2 additional courses of therapy and then receive arsenic trioxide alone twice weekly in the absence of CR, disease progression, or unacceptable toxicity.

After completion of study treatment, patients are followed every 2 months for at least 1 year.

PROJECTED ACCRUAL: A total of 19-41 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndrome or chronic myelomonocytic leukemia
* International Prognostic Scoring System (IPSS) score ≥ intermediate-1

  * Low IPSS score allowed provided patient meets ≥ 1 of the following criteria:

    * Platelet count ≤ 50,000/mm^3
    * Required platelet or packed red cell transfusions within the past 4 weeks
    * Neutropenic (i.e., absolute neutrophil count < 1,000/mm^3) AND has infections requiring antibiotic treatment
* No prior leukemia or refractory anemia with excess blasts in transformation

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 12 weeks

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Baseline QTc < 500 msec
* QTc interval < 460 msec with potassium > 4.0 mEq/L and magnesium > 1.8 mg/L

Immunologic

* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to study drugs
* No ongoing or active infection
* HIV negative

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No other malignancy within the past 12 months

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior administration of any of the following:

  * Interferon
  * Filgrastim (G-CSF), sargramostim (GM-CSF), epoetin alfa, or other hematopoietic cytokines
  * Thalidomide or thalidomide analogs
* No concurrent epoetin alfa

Chemotherapy

* More than 4 weeks since prior chemotherapy
* No prior arsenic trioxide or azacitidine
* No other concurrent chemotherapy

Endocrine therapy

* More than 4 weeks since prior steroids
* No concurrent androgenic steroids

  * Concurrent steroids for adrenal failure or as prophylaxis for nausea allowed

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 4 weeks since prior retinoids
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-04; Primary Completion 2006-08-11 (Actual); Study Completion 2006-08-11 (Actual)

PRIMARY OUTCOMES:
Response rate (overall and confirmed) as measured by International Working Group (IWG) standardized criteria for MDS at day 113 and then every 4 weeks until completion of study treatment

SECONDARY OUTCOMES:
Time to treatment failure as assessed by the Kaplan-Meier method at completion of study treatment
Progression-free survival as assessed by the Kaplan-Meier method at completion of study treatment
Toxicity as assessed by the Kaplan-Meier method and NCI-CTCAE version 3.0 during treatment until 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert K. Stuart, MD, Study Chair — Medical University of South Carolina
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States